CLINICAL TRIAL: NCT03689725
Title: The Effect of Music on Functional Processing and Structural and Functional Development of the Preterm Infant's Brain
Brief Title: The Effect of Music on Preterm Infant's Brain Development
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatric Clinical Research Platform (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SNF 32473B_135817/1
Record Dates: First submitted 2018-08-28; First posted 2018-09-28 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preterm music group (Experimental): Music exposure with headphones
  Interventions: Other: Music
- Preterm control group (No Intervention): headphones without music
- Full-term control group (No Intervention)

INTERVENTIONS:
Other: Music — Music created by A. Vollenweider at least 5 times per week from 33 weeks of gestational age until term-equivalent age
  Arms: Preterm music group

SUMMARY:
Studying the effect of music intervention on preterm infants' brain development by MRI and neurodevelopmental assessments

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants: 33 weeks < gestational age < 37 weeks
* Full-term newborns: 37 weeks gestational age < 42 weeks

Exclusion Criteria:

* Neurological issues or malformations (such as III-IV stade Intraventricular hemorrhage, micro or macrocephaly, hydrocephaly...)
* Because of the high noise caused by nasal continuous positive airway pressure (nCPAP), preterm newborns without at least nCPAP pause before 32 6/7 gestational age will be excluded

Ages: 33 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Estimated)
Dates: Start 2013-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare structural maturation in the three groups using structural MRI and DTI | 40 weeks gestational age
  An MRI will be conducted at term or term equivalent age including structural Magnetic Resonance Imaging and Diffusion Tensor Imaging (DTI) measures.
Compare resting state maturation in the three groups using resting state fMRI | 40 weeks gestational age
  An MRI will be conducted at term or term equivalent age including resting state functional magnetic resonance imaging (fMRI) measures.

SECONDARY OUTCOMES:
Functional responses to known and unknown music in preterm infants with music intervention will be compared to no-intervention groups responses using fMRI | 40 weeks gestational age
  fMRI will be conducted in all three groups at term or term equivalent age
Functional responses to known and unknown music in preterm infants with music intervention will be compared to no-intervention groups responses using EEG | 40 weeks gestational age
  High density Electroencephalography (EEG) will be conducted in all three groups at term or term equivalent age (mismatch negativity, Delta Brushes)
The music intervention effect on cognitive language and motor development at one and two years of age | at 1 and 2 years of age
  Bayley III Cognitive / Language (receptive / expressive) / Motor (fine / gross) Child's performance is compared with norms taken from typically developing children of their age (in months)
The music intervention effect on emotion and temperament at one and two years of age | at 1 and 2 years of age
  LABoratory Temperament Assessment Battery (LabTAB)
  Four episodes:
  * "Puppet Game": Joy (mean of Facial, Vocal, and Bodily responses 0-3); Avoidance (negative motor action 0-3)
  * "Attractive Toy Placed Behind Barrier": Frustration/Anger (0-3); Avoidance (0-3)
  * "Unpredictable Mechanical Toy": Fear (mean of Vocal and Facial responses 0-3) ; Approach (0-3)
  * "Blocks": Attention (mean of Manipulation, Regards, Facial interest 0-3) A higher score indicates more emotional reactivity during a specific emotion-eliciting situation.
The music intervention effect on effortful control at one and two years of age | at 2 years of age
  Effortful control battery Episodes: "Snack Delay", "Wrapped Gift", and "Tower". These episodes evaluate two components of effortful control: delaying (waiting for a pleasant event) twice and suppressing or initiating activity to signal (taking turns), respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Petra S. Hüppi, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sa de Almeida J, Baud O, Fau S, Barcos-Munoz F, Courvoisier S, Lordier L, Lazeyras F, Huppi PS. Music impacts brain cortical microstructural maturation in very preterm infants: A longitudinal diffusion MR imaging study. Dev Cogn Neurosci. 2023 Jun;61:101254. doi: 10.1016/j.dcn.2023.101254. Epub 2023 May 11. PMID 37182337